CLINICAL TRIAL: NCT01985971
Title: F18 EF5 PET/CT Imaging in Patients With Brain Metastases From Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 15910
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Brain Metastases From Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EF5 (Experimental)
  Interventions: Radiation: PET/CT Imaging

INTERVENTIONS:
Radiation: PET/CT Imaging

SUMMARY:
To estimate the presence of hypoxia in individual lesions after radiotherapy in patients with brain metastases from breast cancer as identified by F18 EF5 PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with measurable brain metastases of at least 1 cm in any plane based on anatomic imaging.
* Subjects with prior resection of brain metastases with progressions on brain MRI.
* Histologic confirmation of breast cancer.
* Age of study subject must be > 18 years.
* ECOG Performance Status ≤ 2.
* Ability to undergo brain MR and PET imaging
* Study subjects must have normal organ and marrow function as defined below:

WBC >2,000/mmᶟ, platelets >90,000/mmᶟ, total bilirubin <2.0 mg/dl, creatinine <2.0 mg/dl.

* The effects of EF5 on the developing human fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation (1 month). Should a woman become pregnant pr suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women of childbearing potential will have a urine pregnancy test the day of the F18 -EF5 PET scan prior to the F18 -EF5 injection.
* Ability to understand, participate and provide a documented signed informed consent.
* Subjects who are allergic to gadolinium will have MRI scans without gadolinium contrast.

Exclusion Criteria:

* History of allergic reactions attributed to Flagyl (metronidazole), which has a chemical structure similar to EF5.
* Pregnant women are excluded because EF5 has an unknown risk for adverse events in fetuses and nursing infants secondary the administration of EF5 to the mother. Breastfeeding should be discontinued if EF5 is administered to the mother.
* Subject has any other condition or personal circumstance that, in the judgement of the investigator, might interfere with the collection of complete good quality data.
* Subjects who are unable to provide informed consent.
* Patients with prior whole brain radiotherapy.
* Patients with moderate to severe renal failure, defined as estimated GFR less than 30 ml/Lmin 1.73m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-03; Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilie Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- F18 EF5 PET/CT Imaging: PET/CT Imaging
Period: Overall Study
Arm/Group | F18 EF5 PET/CT Imaging
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- EF5 PET/CT Imaging: PET/CT Imaging
Arm/Group | EF5 PET/CT Imaging
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | EF5 PET/CT Imaging
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Arm/Group | EF5 PET/CT Imaging
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes